CLINICAL TRIAL: NCT07063719
Title: Identification of Cellular Biomarkers of Rare Eye Diseases in Adults
Acronym: REVIBIO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C24-15
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Rare Diseases; Ophthalmology
Keywords: Rare occular disease
MeSH Terms: conditions — Rare Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional interventional research with minimal risks and constraints, national and multi-center clinical study carried out as part of the overall EU project. This WP2 study will be performed in two other countries: Germany (UKK) and Italy (OSR). Each partner will have the responsibility for the clinical study carried out in its country.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): In France, two groups of participants will be recruited (110 participants). 55 of subjects in a control group, will be selected to match the two groups with regard to possible confounding variables, such as gender and age (±5). Patients in the control group will be recruited from the ophthalmology clinics of the Cochin and Necker hospitals, as these patients are already being treated in these hospitals for other pathologies unrelated to rare diseases.
  Interventions: Other: Ophthalmological visit; Other: Questionnaires; Other: Blood sample collection; Other: Impression cytology; Other: Tear fluid
- Patient group (Other): In France, two groups of participants will be recruited (110 participants). 55 subjects with REDs in an experimental group. This group is divided into subgroups. Indeed, 15 patients will be affected by AAK, 5 by NK, 5 by LSCD, 10 by OCP, 5 by Oc GvHD, 10 by EEC and 5 by CNV (the 7 different rare eye diseases)
  Interventions: Other: Ophthalmological visit; Other: Questionnaires; Other: Blood sample collection; Other: Impression cytology; Other: Tear fluid

INTERVENTIONS:
Other: Ophthalmological visit — Uncorrected visual acuity (UCVA), best-corrected visual acuity (BSCVA), corneal topography, corneal pachymetry, ocular surface pictures (to evaluate disease status of the eye with and without fluorecein), Schirmer's test, Corneal esthesiometry, Tear film break-up time test, Intraocular pressure.
  Below is a summary of steps to perform ocular surface pictures of the cornea.
  1. Ensure slit lamp cleaning and appropriate magnification and light settings.
  2. Ensure comfortable positioning of both the operator and the patient.
  3. Examine external orbital structures and adnexa for inflammation, irritation, or lesions.
  4. Examine lids and lashes for abnormalities.
  5. Examine both bulbar and palpebral conjunctiva for signs of irritation and injection.
  6. Examine the cornea for clarity and the presence of any defect.
  7. Examine the anterior chamber depth and evaluate abnormalities that might affect its transparency (blood, purulent material, cells and flare).
  8. Examine the surface of the iris an
Other: Questionnaires — Ocular Surface Disease Index (OSDI) questionnaire, Visual Analog Pain Scale (VAS) questionnaire
Other: Blood sample collection — Blood samples from RED patients or control group are collected in BD Vacutainer K2 EDTA.
Other: Impression cytology — Put one drop of oxybuprocaine hydrochloride 0.4% in patients' eyes and wait 10 seconds. Gently apply both side of one sterile nitrocellulose membrane onto the unexposed bulbar conjunctiva, superotemporally, inferotemporally, superonasally, and inferonasally, for approximately 20 seconds, please, keep the eyes separated.
Other: Tear fluid — One sterile minisponge per eye will be placed over the lids margin at the junction of the lateral and middle thirds of the lower eyelids and kept in place for 2 minutes. During application of sponges the patient needs to look up to facilitate the procedure. To avoid excessive tear reflex, as well as a mild discomfort, it is recommended that patients close their eyes during the collection. Remove sponge using sterile tweezers and put it into empty 0.5mL tube (pierced at the bottom with a sterile needle) placed into another empty 1.5 mL tube and keep it on ice until processing.

SUMMARY:
The cornea is the outermost transparent 'window' of the eye allowing light to enter and serving as the first-line immune and mechanical barrier. It is a complex avascular tissue composed of cells, stem cells, nerves, and collagen layers organized in an exquisite manner to maintain its transparency and self-healing capacity. This delicately balanced interplay of corneal elements is disrupted in rare diseases of the cornea, resulting in non-healing wounds, corneal ulceration, inflammation, new vessel ingrowth (neovascularization), defective innervation, scarring, oedema and loss of transparency. For many Rare Eye Diseases (REDs), drug development has been relatively unsuccessful, delivering few to no new therapies. Current management is often prohibitively expensive, has low efficacy and leads to debilitating side effects. The RESTORE VISION project (https://restorevision-project.eu/) aims to improve eye health by using cutting-edge models for each rare disease to test novel and repurposed compounds (9 in total) and determine drug mechanisms of action, formulating compounds as safe eye drop suspensions, and performing several first-in-human trials of novel therapies. Thes drugs have solid preliminary data showing beneficial effects in restoring the cell physiology, immune, avascular, neural and signaling environment in the cornea.

The current clinical study is part of Work package 2 within the RESTORE VISION EU grant agreement (''Validation of human drug targets of repurposed drugs and novel therapies'') and aims to ascertain the expression levels of genes and proteins and investigate pathways of interest in human tissue and fluid samples of REDs, that are targeted by the proposed experimental/repurposed substances. Therapeutic target gene and/or protein expression will be verified in human blood, tears and conjunctival cells collected from 7 RED patient groups. The RESTORE VISION Consortium know multiple putative genes and proteins involved in the REDs and/or affected by the drugs to be tested in RED models. These will be analyzed in patient samples from the 7 REDs to see if they are 1) expressed at all; 2) differ in expression between patient and control group and 3) are correlated with clinical endpoints and/or symptoms of REDs.

The 7 REDs under investigation are briefly explained as follows:

1. AAK: genetic progressive limbal stem cell degeneration leading to corneal neovascularization, inflammation, recurrent erosions, chronic pain and vision loss.
2. OCP: autoimmune scarring of the conjunctiva leads to deficient wound healing, inflammation, scarring, blindness and pain.
3. EEC Syndrome: Ectodermal Dysplasia causes pathological corneal scarring and blindness.
4. NK: involves a corneal nerve deficit leading to reduction or loss of corneal sensitivity, impaired wound healing, corneal ulceration and loss of vision.
5. LSCD: acquired or hereditary stem cell deficiency inducing epithelial breakdown, neovascularization, scarring and inflammation leading to decreased vision, tearing and pain.
6. oGvHD: a severe side-effect of successful bone-marrow transplantation leads to painful and blinding ocular surface inflammation, neovascularization and delayed wound healing.
7. CN: in high-risk transplantation, pathologic inflammation, corneal blood and lymphatic vessels are key risk factors for high-risk corneal graft failure, leading to graft rejection and blindness.

DETAILED DESCRIPTION:
The expression levels of the genes/proteins that are investigated in this study will be differentially expressed (up/down regulated) between patient and control groups and furthermore there will be associations between the expression levels of these genes/proteins* and clinical endpoints/symptoms in patients with the 7 REDs. The analysis that will be performed in this study will provide key insights into mechanisms of disease in the 7 REDs and the pathways targeted by the RESTORE VISION drugs.

*Restore Vision REDs and gene/protein targets :

Impression cytology :

* For AAK : PAX6, IRS-1, MR, GR, HSD1, HSD2
* For OCP : IRS-1,MR, GR
* For EEC : IRS-1, MR, GR, HSD1, HSD2
* For NK : IRS-1, MR, GR, HSD1, HSD2
* For LSCD : IRS-1, MR, GR, HSD1, HSD2, DCN/LRG-1
* For oGvHD : IRS-1, MR, GR, HSD1, HSD2
* For CN : IRS-1, MR, GR, HSD1, HSD2, DCN/LRG-1

Tear fluid :

* For AKK : PAX6
* For EEC : SPRR1A
* For LSCD :DCN/LRG

ELIGIBILITY:
Inclusion Criteria:

Patient group:

* Women and men with age equal or higher than 18 years (patients planning to conceive may be included in the study)
* Willingness and ability to read and understand the informed consent.
* Diagnosis (including genotype, if needed) of REDs.
* Affiliation with a social security scheme or beneficiary of such a scheme.

RED 1 - AAK Diagnosis criteria

* Compatible slit lamp examination (iris/pupillary abnormalities, with or without corneal opacification, vascularization, cataract, glaucoma). with or without:
* Foveal hypoplasia and optic disc malformations as detected through fundus examination or OCT tomography
* Compatible anterior segment OCT or high-frequency ultrasound biomicroscopy (UBM)
* Positive genetic testing

RED 2 - NK Diagnosis criteria

* Compatible history and slit lamp findings of one of the three stages of the Mackie classification (I - punctate keratopathy; II - persistent epithelial defect; III - stromal involvement)
* Reduced/absent corneal sensitivity
* Exclusion of infectious or toxic etiologies with or without:
* confocal microscopy findings

RED 3 - LSCD Diagnosis criteria

* Compatible history and slit lamp examination (e.g. corneal conjunctivalization with persistent epithelial defects, loss of limbal anatomy or irregular staining with fluorescein) with or without:
* confocal microscopy findings

RED 4 - OCP Diagnosis criteria

* Compatible slit lamp examination
* Exclusion of infectious or toxic etiologies with or without:
* conjunctival /oral biopsy with characteristic mucous pemphigoid findings

RED 5 - OC GVHD Diagnosis criteria • Compatible history and slit lamp examination consistent with one of 4 grades of ocular GVHD (1 - conjunctival hyperemia, 2 - fibrovascular changes <25% of palpebral conjunctiva, 3 - fibrovascular changes >25%, 4 - >75% or cicatricial entropion)

RED 6 - EEC Diagnosis criteria

* Compatible slit lamp examination
* Compatible systemic findings with or without:
* Positive genetic testing

RED 7- CNV Diagnosis criteria

* Compatible slit lamp examination of corneal stromal neovascularization (1-4 quadrants)
* Exclusion of infectious or toxic etiologies with or without:
* confocal microscopy findings

Control group:

* Women and men with age equal or higher than 18 years (patients planning to conceive may be included in the study).
* Willingness and ability to read and understand the informed consent.
* Non-diagnosis of REDs.
* Affiliation with a social security scheme of beneficiary of such a scheme.

Exclusion Criteria:

Patient group:

* Pregnancy, breastfeeding (in case any stress was caused to the woman by the biological sampling).
* Descemetocele/impending corneal perforation.
* Recent (less than 3 months) ocular surgery.
* Recent (less than 1 month) change in topical medications type and frequency of the ocular pathology.
* Persons subject to a legal protection measure (under guardianship, curatorship or safeguard of justice)

Control group:

* Pregnancy, breastfeeding.
* Active ocular infection.
* Descemetocele/impending corneal perforation.
* Recent (less than 3 months) ocular surgery.
* Recent (less than 1 month) change in topical medications type and frequency of the ocular pathology.
* Persons subject to a legal protection measure. (under guardianship, curatorship or safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
The expression levels of the genes and proteins | At the inclusion visit
  The primary endpoint will be the expression levels of the genes and proteins listed in the Study description. These genes and proteins are expected to be differentially expressed (upregulated or down regulated) compared to the control group. The investigators will arbitrarily set at 1 the target level in the control group and the RED group will be expressed in relation to the control group.
  While sample collection occurs in 4 Clinical centers (2 in Inserm, France, 1 in Klinikum der Universitaet zu Koeln (UKK, Germany) and 1 in San Raffaele Hospital OSR, Italy), following any initial required processing all samples will be shipped to OSR in Italy who will perform the qPCR, Elisa and/or Mass Spectrometry analysis. Laboratory tests (qPCR, Elisa and/or Mass Spectrometry) will be performed at the Eye Repair lab of the Department of Neuroscience at IRCCS at OSR.

SECONDARY OUTCOMES:
The expression levels of the genes and proteins | At the inclusion visit
  The secondary endpoint will again be expression levels of the genes and proteins listed in the study description, however then these genes and protein expression levels will be analyzed statistically to see if there are correlations with the clinical measurements taken in this study (pictures, health questionnaires, uncorrected visual acuity, best spectacle corrected visual acuity, corneal topography, corneal pachymetry and the slit lamp pictures acquired during the ophthalmologic exam).
  The measurement of the secondary endpoints will be performed using the same timepoint and techniques as are planned to be used for measurement of the primary endpoints which will be combined with statistical analysis to identify any correlations between gene/protein expression levels in RED patients and controls and the clinical measurements taken in this study.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Universitaire Cochin, APHP, Paris
  - Hôpital Universitaire Necker Enfants malades, APHP, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stachon T, Fecher-Trost C, Latta L, Yapar D, Fries FN, Meyer MR, Kasmann-Kellner B, Seitz B, Szentmary N. Protein profiling of conjunctival impression cytology samples of aniridia subjects. Acta Ophthalmol. 2024 Jun;102(4):e635-e645. doi: 10.1111/aos.16614. Epub 2023 Dec 21. PMID 38130099
- [Background] Lasagni Vitar RM, Bonelli F, Atay A, Triani F, Fonteyne P, Di Simone E, Rama P, Mondino A, Ferrari G. Topical neurokinin-1 receptor antagonist Fosaprepitant ameliorates ocular graft-versus-host disease in a preclinical mouse model. Exp Eye Res. 2021 Nov;212:108825. doi: 10.1016/j.exer.2021.108825. Epub 2021 Nov 3. PMID 34740637